CLINICAL TRIAL: NCT07281508
Title: Transtympanic Sodium Thiosulfate to Prevent Cisplatin-related Hearing Loss A Randomized Controlled Multicenter Phase III Trial; The SOUND Trial
Brief Title: Transtympanic STS Against Cisplatin-induced SNHL: the SOUND Trial
Acronym: SOUND
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: M21STS
Record Dates: First submitted 2023-06-27; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Cisplatin-related Hearing Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transtympanic sodium thiosulphate (STS) 0.1M/0,5% hyaluronate (Experimental): One ear of a patient: The transtympanic sodium thiosulphate is administered into one ear of a patient. The intervention takes place within 3 hours before each cisplatin course. The intervention takes place 3 to 7 times, depending on the cisplatin schedule
  Interventions: Drug: Transtympanic sodium thiosulphate (STS) 0.1M/0,5% hyaluronate
- Untreated ear (No Intervention): The other ear of the same patient is left untreated

INTERVENTIONS:
Drug: Transtympanic sodium thiosulphate (STS) 0.1M/0,5% hyaluronate — The transtympanic injection gel is composed of the following components:
  * Sodium Thiosulfate 250mg/mL, 10mL for injection (STS)
  * BiolevoxTM HA 2,2%, 2mL, pre-filled syringe for intraarticular injection (HYA)
  * Sterile Phosphate-buffered Sodium Chloride, 500mL (PBS)
  Arms: Transtympanic sodium thiosulphate (STS) 0.1M/0,5% hyaluronate

SUMMARY:
The goal of this clinical trial is to learn if transtympanic sodium thiosulfate (STS) injections can prevent hearing loss caused by cisplatin chemotherapy in adults with head and neck cancer. The main question it aims to answer is:

Researchers will compare the ear treated with STS gel to the untreated ear within the same patient to see if STS prevents hearing loss.

Participants will:

1. Receive STS gel injections into the middle ear of one ear (randomized) within 3 hours before each cisplatin infusion (3-7 injections per patient).
2. Undergo hearing tests at baseline and 2-4 months after the last cisplatin treatment.
3. Complete questionnaires about hearing and tinnitus at baseline and 2-4 months after treatment.

DETAILED DESCRIPTION:
Trial design:

This study is an investigator-initiated randomized controlled multicenter phase III trial. Patient accrual and treatment (treatment and hearing analysis will take 22 weeks per patient) will start in 2025 and will be completed in 2028. Afterwards, the patients will have a routine follow-up for a median of 2 years to collect necessary survival data (2025-2030).

Trial population:

A hundred patients with solid head and neck malignancies who are treated with ≥ 200 mg/m2 cisplatin will be included. To be eligible for participation, patients must be 18 years or older. Study participation is not possible if more than 30 gray radiotherapy is applied to the inner ear, asymmetric hearing loss or more than 40 dB hearing loss is detected before start of treatment, known hypersensitivity to STS injections, and/or if patients have ear conditions that prevent middle ear injections from being administered properly.

Interventions:

Patients will be treated with an STS injection in one ear and no treatment in the contralateral ear. The ear to be treated with STS gel will be determined by randomization. The hearing of the treated ear will then be compared with the untreated ear. The audiometrist who conducts the hearing test will not know which ear has been treated with sodium thiosulfate. Hence, the design of this trial takes advantage of the fact that every patient has two ears, and offers the unique concept of having a randomized controlled comparison of platinum-induced hearing loss of the treated versus the untreated ear within individual patients. This results in the advantage that during the analysis of the results differences between patients are eliminated. The STS gel will be injected into the middle ear within three hours before each cisplatin infusion (range 3-7 injections per patient) into one ear, the other ear will be left untreated. Hearing tests will be conducted at baseline (before the first cisplatin therapy) and 3 months (range 2 - 4) after the last cisplatin infusion. Questionnaires will be filled in to document hearing-related complaints at baseline and 3 months (range 2 - 4) after the last cisplatin treatment. For the survival analysis on a median of 1 and 2 years after treatment, survival data will be collected from the patient's medical records. These data will be compared to similar patients from historical data. In a pilot of 10 patients in the LUMC vestibular testing will be performed at baseline and 6 weeks after the last cisplatin infusion.

Ethical considerations relating to the clinical trial including the expected benefit to the individual subject or group of patients represented by the trial subjects as well as the nature and extent of burden and risks:

Based on the results of our successfully completed phase I study, we expect that 30-50% of patients will experience a noticeable difference between the STS-treated and untreated ear (2). The STS injections in the middle ear carry small risk. Our phase 1 study has shown that administrations of sodium thiosulfate are safe. The possible risks/side effects of the injections are pain, temporary fullness in the ear, temporary dizziness, and temporary decreased hearing. There is also a very small (<1%) risk of permanent perforation of the eardrum. The injections will be given before every cisplatin treatment because sodium thiosulfate remains available in the middle and inner ear for only a temporary period. The METC does not agree with the use of a placebo control, as the risk of a complication (albeit small) is not acceptable. The current standard of care is 'no treatment' and the audiogram provides a sufficiently objective measurement. Therefore, the study design is changed to a non-placebo randomised controlled trial and only the audiometrist is blinded.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological proof of solid head and neck malignancies with an indication for treatment with cisplatin in a cumulative dose of ≥ 200mg/m2 given in a weekly schedule of 7 times 40 mg/m2 or a 3-weekly schedule of 3 times 100 mg/m2
* Treatment with high-dose cisplatin (cumulative dose ≥ 200mg/m2) of maximum 7 cycles
* Able and willing to give written informed consent;
* WHO performance status of 0, 1 or 2;
* Age older than 18 years.

Exclusion Criteria:

* Asymmetric hearing capacity (SNHL) prior to treatment, defined as a difference between both ears in hearing capacity of ≥ 10 dB averaged over 3 adjacent frequencies in the range of 0.5 to 12.5 kHz (i.e. 0.5, 1, 2, 4, 8, 10 and 12.5 kHz).
* Baseline hearing: more than 40 dB SNHL at PTA 1-2-4 kHz (in one or both ears)
* A planned radiation dose of > 30 Gy to the cochlea (8);
* Known hypersensitivity to STS-containing HYA gel formulation;
* Any condition that would, according to the investigator's judgement, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures;
* Otologic pathology that hampers the transtympanically applied STS gel to diffuse through the round window, e.g. otosclerosis, a narrow ear canal, otitis media with effusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2030-03-23 (Estimated); Study Completion 2030-03-23 (Estimated)

PRIMARY OUTCOMES:
The efficacy (clinically relevant benefit) of transtympanic STS 0.1M/0.5 HYA against platinum-related ototoxicity. | Baseline and 2-4 months after last cycle of chemotherapy
  The percent of patients with a clinically relevant benefit of transtympanic STS injection against CIHL, defined as the change in the threshold between baseline and 3 months after treatment differs by ≥ 10 dB at any three adjacent frequencies from 0.5 to 16 kHz in favour of the STS treated ear.

SECONDARY OUTCOMES:
The superiority of STS versus untreated ear with regard to hearing capacity based on audiometry. | Baseline and 2-4 months after last cycle of chemotherapy
  Mean difference between STS- and untreated ears in threshold shift (post-treatment minus baseline hearing, in a continuous scale) at sensorineural pure tone averages (PTA) 1-2-4 kHz and 8-10-12.5 kHz in dB.
The superiority of STS versus untreated ear with regard to hearing loss based on American Speech-Language-Hearing Association criteria (ASHA). | Baseline and 2-4 months after last cycle of chemotherapy
  The difference in sensorineural hearing loss between STS- and placebo-treated ears based on the ASHA criteria:
  * Grade A: threshold shift ≥ 20 dB at any one test frequency;
  * Grade B: threshold shift ≥ 10 dB at 2 consecutive frequencies;
  * Grade C: loss of response at three consecutive test frequencies where responses were previously obtained (this refers specifically to the highest frequencies tested, where earlier responses are obtained close to the limits of the audiometric output and later responses cannot be obtained at the limits of the audiometer).
The superiority of STS versus untreated ear with regard to hearing loss based on TUNE criteria. | Baseline and 2-4 months after last cycle of chemotherapy
  The difference in sensorineural hearing loss between STS- and placebo-treated ears based on the TUNE criteria:
  * Grade 0: No hearing loss
  * Grade 1a: threshold shift ≥ 10dB at PTA 8-10-12.5 kHz OR subjective hearing changes without threshold shift
  * Grade 1b: threshold shift ≥ 10dB at PTA 1-2-4 kHz
  * Grade 2a: threshold shift ≥ 20dB at PTA 8-10-12.5 kHz
  * Grade 2b: threshold shift ≥ 20dB at PTA 1-2-4 kHz
  * Grade 3: Hearing level ≥ 35dB HL at PTA 1-2-4 kHz de novo
  * Grade 4: Hearing level ≥ 70dB HL at PTA 1-2-4 kHz de novo
The superiority of STS versus placebo-treated ear with regard to hearing loss based on the Common Terminology Criteria for Adverse Eventes (CTCAE) criteria. | Baseline and 2-4 months after last cycle of chemotherapy.
  The difference in sensorineural hearing loss between the STS- and placebo treated ears based on the CTCAE criteria (40):
  * Grade 1: threshold shift of 15 - 25 dB averaged at 2 contiguous test frequencies in at least one ear OR subjective change in hearing in the absence of documented hearing loss;
  * Grade 2: threshold shift of > 25 dB averaged at 2 contiguous test frequencies in at least one ear;
  * Grade 3: threshold shift of > 25 dB averaged at 3 contiguous test frequencies in at least one ear OR hearing aid or intervention indicated
  * Grade 4: Decrease in hearing to profound bilateral loss (absolute threshold > 80 dB HL at 2 kHz and above); non-serviceable hearing
Survival | 1 and 2 years after the start of treatment.
  Disease-specific survival, recurrence-free and overall survival measured at median 1 and 2 years after the start of treatment.
Quality of life/Patient-related outcome measures (PROM). Subjective hearing loss after platinum treatment. | Baseline and 2-4 months after last cycle of chemotherapy
  For the evaluation of patient reported outcome measurements concerning hearing loss, we use the following questionnaire:
  Speech, Spatial and Qualities of Hearing scale (SSQ) 12. This questionnaire
  Each item on the questionnaire (12 questions) shows a ruler with a 10-point scale on which the responders can rate themselves. The left hand-end, or lowest grade, of the ruler represents the complete inability or complete absence of a quality, whereas the right hand represents the complete ability or complete presence of a quality.
Quality of life/Patient-related outcome measures (PROM). Subjective tinnitus after platinum treatment. | Baseline and 2-4 months after last cycle of chemotherapy
  For the evaluation of patient reported outcome measurements concerning potential development of tinnitus, we use the following questionnaire:
  Tinnitus Handicap Inventory (THI)-12.
  The THI (12 questions) scores different degrees of severity of tinnitus, i.e. slight, mild, moderate and severe, which depends on the score obtained from the responder's answers on the questionnaire.

OTHER OUTCOMES:
Cisplatin-related vestibulotoxicity | Baseline and 6 weeks after last cycle of chemotherapy.
  To assess cisplatin related vestibulotoxicity based on vestibular testing (V-HIT) at baseline and 6 weeks post-treatment in the STS-treated ear versus untreated ear and to evaluate the preventive effect of transtympanic STS injections on cisplatin-related vestibulotoxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Lotje Zuur, Prof. Dr., Principal Investigator — AVL
Locations (5):
- Netherlands (5):
  - Antoni van Leeuwenhoek, Amsterdam, North Holland
  - Leiden University Medical Center, Leiden, South Holland
  - Erasmus Universitair Medisch Centrum Rotterdam, Rotterdam, South Holland
  - University Medical Center Utrecht, Utrecht, Utrecht
  - Stichting Radboud University Medical Center, Nijmegen

IPD SHARING:
Plan to Share IPD: Yes
For future research, other than defined in the protocol, a request for use of the data has to be performed. Only with ethical clearance by the METC or IRB NKI, an investigator will be allowed to use this data.